CLINICAL TRIAL: NCT07385703
Title: A Randomized, Open-Label, Multicenter Phase III Study of Tecotabart Vedotin Plus Tislelizumab Versus Tislelizumab Plus Chemotherapy as First-Line Treatment in Patients With CLDN18.2-Positive, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Clinical Study on the Efficacy and Safety of LM-302 Injection Combined With Tislelizumab and Tislelizumab Combined Chemotherapy for the Treatment of Gastric or Gastroesophageal Junction Adenocarcinoma.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM302-03-201
Record Dates: First submitted 2026-01-25; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — tislelizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-302 Injection+Tislelizumab (Experimental): LM-302 Injection combined with Tislelizumab, 14days as a treatment cycle.
  Interventions: Drug: LM-302 Injection; Drug: Tislelizumab
- Tislelizumab + oxaliplatin Injection +Capecitabine Tablets (Active Comparator): Tislelizumab combined with oxaliplatin and capecitabine tablets, 21days as a treatment cycle.
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin Injection; Drug: Capecitabine Tablets

INTERVENTIONS:
Drug: LM-302 Injection — The LM-302 injection is an ADC drug targeting CLDN18.2.
  Arms: LM-302 Injection+Tislelizumab
Drug: Tislelizumab — Tislelizumab is a humanized monoclonal antibody targeting programmed cell death receptor-1 (PD-1).
Drug: Oxaliplatin Injection — Oxaliplatin injection is a platinum-based antitumor drug.
  Arms: Tislelizumab + oxaliplatin Injection +Capecitabine Tablets
Drug: Capecitabine Tablets — Capecitabine tablets belong to the fluorouracil-class prodrugs.
  Arms: Tislelizumab + oxaliplatin Injection +Capecitabine Tablets

SUMMARY:
This study primarily evaluates the efficacy and safety of the LM-302 plus tislelizumab regimen versus tislelizumab plus chemotherapy in the treatment of previously untreated locally advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma patients with CLDN18.2 positivity.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with the study's visit schedule, treatment plan, laboratory tests, and other research procedures.
* Age ≥ 18 years.
* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction.
* For locally advanced unresectable or metastatic adenocarcinoma of the stomach or gastroesophageal junction that has not previously received any systemic treatment:

  * Patients who have previously received radical neoadjuvant chemotherapy or adjuvant chemotherapy (radiotherapy) based on a platinum-based combination chemotherapy regimen and have not developed distant metastasis or local recurrence within 6 months after completion of treatment can be included.
  * The calculation of a 6-month interval is defined as recurrence within the same date range after 6 months. For example, if the end date of the last treatment is January 1, the 6-month period from that date refers to January 1 to July 1 (including July 1). Alternatively, if the end date of the last treatment is August 31, the 6-month period from that date refers to August 31 to February 28 (or February 29 in leap years).
* Archived specimens or fresh tumor tissue specimens from ≤3 years ago must be provided for CLDN18.2 and PD-L1 testing (PD-L1 results are not a condition for enrollment). When multiple samples are present, the most recent accessible and qualified sample must be provided. After confirmation by the central laboratory, tumor tissue with positive CLDN18.2 expression is defined as ≥25% tumor cell membrane staining intensity 2+ & 3+. For patients who have previously received radical neoadjuvant chemotherapy or adjuvant chemotherapy (radiotherapy) based on platinum-containing combination chemotherapy regimens, newly obtained tissue from recurrent or metastatic lesions must be provided for CLDN18.2 and PD-L1 testing.
* A negative report on the expression detection of human epidermal growth factor receptor-2 (HER2) in tumor tissue must be provided. The definition of HER2 negative expression is ImmunoHistoChemistry (IHC) score 0/1+, IHC score 2+, and fluorescence in situ hybridization (FISH) negative.
* According to the RECIST 1.1 evaluation criteria, there must be at least one measurable lesion.
* Expected survival duration ≥ 3 months.
* According to the Eastern Cooperative Oncology Group (ECOG) standards, the physical performance status score is 0 or 1.
* Good organ function: a. Bone marrow reserve: Platelets (PLT) ≥ 100×10^9/L, absolute neutrophil count (ANC) ≥ 1.5×10^9/L, Hemoglobin (Hb) ≥ 90 g/L (no blood transfusion or supportive treatment such as colony-stimulating factors within 14 days prior to hematology parameter examination during the screening period); b. Coagulation function: International normalized ratio (INR) ≤ 1.5, Activated partial thromboplastin time (APTT) ≤ 1.5×upper limit of normal (ULN); c. Liver function: Total bilirubin ≤ 1.5×ULN, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase (ALP) ≤ 2.5×ULN (if there is liver metastasis, then ALT and AST ≤ 5×ULN) and Albumin (ALB) ≥ 30 g/L; d. Renal function: Creatinine clearance rate ≥ 50 mL/min (calculated according to the Cockcroft-Gault formula); e. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; QT interval (QTcF) ≤ 470 ms for females and ≤ 450 ms for males.
* Women of childbearing age must have a negative blood pregnancy test within 7 days before administration; any fertile male and female subjects must agree to use highly effective contraception throughout the study medication period and for 7 months after the last dose of the study. Males must agree to refrain from donating sperm during the study period and for 7 months after the last dose of the study. Females must agree to refrain from breastfeeding during the study period.

Exclusion Criteria:

* Other pathological types confirmed by histopathology, such as squamous cell carcinoma, sarcoma, or undifferentiated carcinoma.
* There are gastric cancer lesions confirmed by imaging that are accompanied by cavities or necrosis, and are closely related to major blood vessels, and are assessed by the researchers as posing a high risk of major bleeding.
* Patients with known central nervous system (CNS) metastases. Patients with non-meningeal, midbrain, pontine, or spinal cord metastases who are judged by the investigator to have stable brain metastases can be enrolled. Stable brain metastases are defined as patients whose brain metastases have undergone treatment and the condition of the metastases has stabilized (brain imaging examination at least 28 days before randomization shows stable lesions, no neurological symptoms, and no immediate need for local or systemic treatment within 14 days before randomization), with no evidence of new or previously existing brain metastases enlarging.
* Clinically uncontrollable third-space effusion, such as moderate or greater volume, requiring long-term catheterization, previous history of intestinal obstruction or paralysis, compartmented ascites, undergoing or planning to undergo local treatment (including drainage, peritoneal shunt, or cell-free concentrated ascites reinfusion therapy) within 14 days prior to screening, or significant increase within 2 weeks after local treatment, meeting any of the above criteria or deemed unsuitable for enrollment by the investigator.
* Patients with symptomatic spinal cord compression, or those who are expected to develop symptoms of spinal cord compression if left untreated; or for patients with previously diagnosed and treated spinal cord compression, there is no evidence indicating that the disease was clinically stable for ≥4 weeks before the first study drug administration; except for patients with asymptomatic spinal cord compression indicated by imaging, who are assessed as stable by a specialist and do not require treatment for spinal cord compression at this time.
* Accompanied by severe peritoneal metastasis, the main manifestations are: clinically significant intestinal obstruction; barium enema indicating small intestinal stenosis.
* History of gastrointestinal perforation or gastrointestinal fistula within the previous 6 months. If the perforation or fistula has been treated through resection or repair surgery, and the condition is assessed by the investigator as having been cured or controlled, participation in the study is permissible.
* Poorly controlled tumor-related pain:

  * For patients requiring analgesic treatment, a stable dosage of treatment must be established before participating in the study.
  * Symptomatic lesions suitable for palliative radiotherapy (such as bone metastasis or metastasis causing nerve damage) should be treated before enrollment.
  * Before enrollment, if appropriate, consideration should be given to local treatment for asymptomatic metastatic lesions that may lead to functional deficits or intractable pain due to further growth (e.g., epidural metastasis not currently associated with spinal cord compression).
* Patients with a body weight of less than 35kg or a body weight loss of more than 10% within 2 months prior to signing the informed consent form.

Exclusion criteria for comorbidities or concomitant conditions:

* History of malignancy other than Gastric Cancer (GC)/GastroEsophageal Junction adenocarcinoma (GEJ) adenocarcinoma within 2 years prior to randomization, with the following exceptions: basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, squamous cell carcinoma of the skin, etc., which have been completely cured and treated.
* History of autoimmune diseases, including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. The following conditions are excluded: • Subjects with autoimmune-related hypothyroidism who are receiving stable-dose thyroid hormone replacement therapy.

  * Subjects with type 1 diabetes who are well-controlled under a stable insulin treatment regimen.
  * Only subjects with skin autoimmune diseases that do not require systemic treatment (such as vitiligo, alopecia, psoriasis, or eczema).
  * Subjects who have recovered from childhood asthma and do not require any intervention in adulthood.
  * Subjects whose relevant diseases, as assessed by the researchers, are unlikely to recur without external triggers.
* Patients who have previously undergone allogeneic bone marrow transplantation or solid organ transplantation.
* Patients with a history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

  * Severe cardiac rhythm or conduction abnormalities, such as arrhythmias requiring clinical intervention, second- or third-degree atrioventricular block, left bundle branch block, prolonged QRS complex, etc.;
  * Patients with thromboembolic events requiring therapeutic anticoagulation, or those with venous filters;
  * Patients with heart failure of New York Heart Association (NYHA) class III or IV;
  * Patients who have experienced acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other cardiovascular and cerebrovascular events of grade 3 or above within the previous 6 months prior to randomization.
  * Have a history of myocarditis or cardiomyopathy.
* For individuals infected with human immunodeficiency virus (HIV) and those with active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, the following conditions are allowed for enrollment: • Patients who are HBsAg positive, with or without HBcAb positivity, and have HBV DNA < 500 IU/mL or below the lower limit of the reference value set by the research center, and who, based on clinical treatment, manifestations, and other factors, are judged by the investigator to have no active infection; • Patients who are HCV antibody positive but HCV RNA negative.
* Subjects with known active syphilis infection.
* Individuals who are unable to control themselves or have severe illnesses, including but not limited to active infections requiring systemic antibiotic treatment within 2 weeks before the first dose, and interstitial pneumonia/lung disease requiring intervention during screening.
* Subjects with known active tuberculosis. For patients suspected of having active tuberculosis, a comprehensive evaluation should be conducted based on chest imaging, sputum smear/culture, or molecular testing results, as well as clinical symptoms and signs, to make a definitive diagnosis.
* Currently present peripheral sensory or motor neuropathy of ≥ grade 2.
* Subjects who received systemic corticosteroids (>10mg/d prednisone equivalent) or other systemic immunosuppressants (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor drugs [anti-Tumor Necrosis Factor (TNF)] within 2 weeks prior to the first study drug administration.

  * Topical, ocular, intra-articular, intranasal, and inhaled corticosteroids are allowed;
  * Patients receiving acute low-dose systemic immunosuppressive drugs (e.g., single-dose dexamethasone for nausea);
  * Patients requiring baseline and subsequent MRI/CT tumor assessments who have previously experienced allergic reactions to intravenous contrast agents may receive prophylactic steroids;
  * Inhaled corticosteroids are allowed for the treatment of chronic obstructive pulmonary disease, hydrocortisone for the treatment of orthostatic hypotension, and low-dose corticosteroid hormone maintenance therapy for adrenal insufficiency.
* There are factors that affect the application and absorption of oral medications, such as dysphagia, clinically uncontrollable persistent and recurrent vomiting (such as caused by gastric outlet obstruction), intestinal obstruction, and chronic diarrhea. 21. Within 28 days before randomization, there was uncontrollable/severe gastrointestinal bleeding, active peptic ulcer, or active gastrointestinal inflammation/infectious diseases (such as active diverticulitis, abdominal abscess). Subjects who have not undergone radical surgical resection of the primary lesion must undergo fecal occult blood testing before enrollment. If the result is positive, further evaluation, including but not limited to gastroscopy, is required before medication administration to confirm the presence of active bleeding from the lesion and assess the risk of bleeding.
* The adverse reactions from previous anti-tumor treatment within the 14 days prior to randomization have not yet recovered to a level of ≤ grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) v6.0 grading system (excluding toxicities that the investigator deems to pose no safety risk, are asymptomatic, or are controllable with stable medication, such as hair loss, long-term toxicity caused by radiotherapy, and other toxicities that are ≤ grade 2).
* Have a history of allergy to LM-302, Ticagrelor, any control drug, or its excipients.
* Individuals with known mental illnesses or disorders that may affect trial compliance.

Exclusion criteria related to drug treatment:

* Within 28 days prior to randomization, the subject is currently participating or has previously participated in any investigational drug study, or has used an investigational device within 28 days. Subjects who have entered the follow-up period of an investigational drug study and have not used the investigational drug for ≥28 days since the last use may meet the inclusion criteria for this study.
* Previously received targeted therapy targeting CLDN18.2, such as antibody-drug conjugate (ADC) therapy, antibody therapy, and chimeric antigen receptor T-cell (CAR-T) therapy; previously received ADC therapy using small molecule toxin Monomethyl auristatin E (MMAE).
* Subjects who have received palliative local treatment (such as radiotherapy or surgery) for non-target lesions within 2 weeks prior to the first dose, or who have previously received radiotherapy for locally advanced unresectable or metastatic gastric cancer or GEJ adenocarcinoma and have not recovered from toxicity within 2 weeks prior to randomization.
* Within the first 2 weeks before randomization, patients received systemic treatment with traditional Chinese patent medicines and simple preparations with anti-tumor indications, or with Chinese herbal medicine, or with drugs with immune regulatory effects (including thymosin, interferon, interleukin, etc.).
* Having undergone or planning to undergo major surgery or interventional therapy (excluding tumor biopsy, puncture, etc.) within the 28 days prior to randomization or during the study period.
* Use of strong inhibitors/strong inducers of CYP3A4 within 14 days before randomization;
* Vaccination with any live vaccine or attenuated live vaccine within 28 days before randomization.
* Other situations where the researcher deems it inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1.5 years
  To compare the progression-free survival (PFS) of patients with locally advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma who were previously untreated and had a PD-L1-positive status (CPS≥1) and high CLDN18.2 expression (≥75% 2+&3+) with the LM-302 plus tislelizumab regimen versus the tislelizumab plus chemotherapy regimen in the LM-302 plus tislelizumab group and in all randomized populations. The PFS was assessed using blind independent central review (BICR) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST1.1) criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | During the study period (Baseline up to two years)
  The preriod from the first use of the drug to death from all causes. For subjects who are still alive at the last follow-up, the OS will be counted as data censored based on the last follow-up. For subjects who are lost follow-up, the OS will be counted as data cesored based on the last confirmed survival time before being lost to follow-up.
Progression-free survival (PFS) assessed by Investigator | During the study period (Baseline up to two years)
  The period from the first use of the drug to disease progression or death (whichever occurs first).
Objective Response Rate (ORR) | During the study period (Baseline up to two years)
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first).
Disease Control Rate (DCR) | During the study period (Baseline up to two years)
  Proportion of subjects whose tumors shrink or remain stable for a certain period, including complete remission (CR), partial remission (PR) and stable disease (SD).
Objective response rates (ORR) | During the study period (Baseline up to two years)
  Proportion of patients whose tumors shrank by a certain amount and remained for a certain period of time, including complete response (CR) and partial response (PR) cases.
Number of subjtecs with incidence of adverse events | During the study period (Baseline up to two years)
  Number of subjtecs with incidence of adverse events: Occurrence of all adverse events (AE), serious adverse events (SAE), and treatment-related adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Locations (104):
- China (104):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital (The First Affiliated Hospital of China University of Science and Technology), Hefei, Anhui
  - The Second Hospital Of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital Of Wannan Medical College, Wuhu, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Lu He Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Gaobo Hospital Co., Ltd., Beijing, Beijing Municipality
  - Beijing Tsinghua changgung Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital Of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong provincial people's hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shantou University Medical College Affiliated Tumor Hospital, Shantou, Guangdong
  - Guigang City People's Hospital, Guigang, Guangxi
  - Guangxi Medical University Afiliated Tomor Hospital, Nanning, Guangxi
  - The People's Hospital of Guizhou Province, Guiyang, Guizhou
  - The Second Affiliated Hospital Of Zunyi Medical University, Zunyi, Guizhou
  - Hainan general hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiamusi Tuberculosis Hospital (Jiamusi Cancer Hospital), Jiamusi, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - The First Affiliated Hospital Of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - The First affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Tongji Hospital Tongji Medical College Of Hust, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Peking University Cancer Hospital Inner Mongolia Hospita, Hohhot, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First People's Hospital Of Changzhou, Changzhou, Jiangsu
  - Jiangsu Provincial Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Fourth Affiliated Hospital Of Soochow University (SuZhou Du Shu Lake Hospital), Suzhou, Jiangsu
  - Xuzhou central hospital, Xuzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Yangzhou Univrtsity, Yangzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Nanchang University First Affiliated Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital Of Nangchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital Of Dalian University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - QinghaiI University Affiliated Hospital, Xining, Qinghai
  - Baoji Central Hospital, Baoji, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital Of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute, Shandong Cancer Hospital), Jinan, Shandong
  - Jinan Central Hospital (City level), Jinan, Shandong
  - Affiliated Hospital Of Ji Ning Medical University, Jining, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Qingdao Municipal Hospital (Group), Qingdao, Shandong
  - Weifang Yidu Central Hospital, Weifang, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - ZhongShan Hospital, Shanghai, Shanghai Municipality
  - Shanghai GoBroad Cancer Hospital China Pharmaceutical University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Chang zhi People's Hospital, Changzhi, Shanxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - First Hospital Of Shan Xi Medical University, Taiyuan, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Sichuan Academy of Medical Science&Sichuan Provincial People' Hospital, Chengdu, Sichuan
  - Sichuan Provincial Cancer Hospital, Chengdu, Sichuan
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lishui Central Hospitall, Lishui, Zhejiang
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang